CLINICAL TRIAL: NCT04828148
Title: Incidence of Infection and Mortality by COVID-19 in Specialists in Mexico: A Cross-sectional Study
Brief Title: Incidence of Infection and Mortality by COVID-19 in Specialists
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal investigator, Instituto Mexicano del Seguro Social
Other Study IDs: Mortality Physicians
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Covid19; Health Care Associated Infection; Infection, Coronavirus; Death
MeSH Terms: conditions — COVID-19; Cross Infection; Coronavirus Infections; Death | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Survey — An online survey made by the authors was used, which is comprised of a total of 48 questions where different types of information are distinguished regarding the participant who is answering it such as age, gender, medical degree, comorbidities if during the pandemic they have been in contact with patients suspected or confirmed of COVID-19 infection if they have been infected by COVID-19 and the outcome of this infection. It also refers to whether they know doctors in the same specialty or others who have died from COVID-19 infection.

SUMMARY:
In this current study the researchers aim to identify the total number of infections and deaths due to COVID-19 and distinguish which are the risk factors most related to COVID-19 infections and deaths in medical personnel in Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Active physicians and medical students who have had contact with patients infected by COVID-19
* Active physicians and medical students who have been infected by COVID-19

Exclusion Criteria:

* Members of the general population
* Inactive physicians or medical students
* Incomplete surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active physicians and medical students who have had contact with COVID-19 patients.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of mortality in physicians due to COVID-19 | Baseline
  An online survey made by the authors was used, which is comprised of a total of 48 questions where different types of information are distinguished regarding the participant who is answering if during the pandemic they refers to whether they know doctors in the same specialty or others who have died from COVID-19 infection.
Incidence of infection in physicians due to COVID-19 | Baseline
  An online survey made by the authors was used, which is comprised of a total of 48 questions where different types of information are distinguished regarding the participant who is answering if during the pandemic they have been in contact with patients suspected or confirmed of COVID-19 infection if they have been infected by COVID-19 and the outcome of this infection.

SECONDARY OUTCOMES:
Physician´s Risk factors of contagion such as age, gender, medical degree, and comorbidities | Baseline
  An online survey made by the authors was used, which is comprised of a total of 48 questions where different types of information are distinguished regarding the participant who is answering it such as age, gender, medical degree, comorbidities, and the association with the severity of the infection by COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Nacional de Occidente, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No